CLINICAL TRIAL: NCT03857711
Title: Multicenter Randomized Clinical Trial PULVAB (Prophylactic Pulmonary Veins Ablation)
Brief Title: Randomized Clinical Trial PULVAB (Prophylactic Pulmonary Veins Ablation)
Acronym: PULVAB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center of Surgery, Russia (Other Government)
Collaborators: Federal Centre of High Medical Technologies of the RF Ministry of Public Health, Kaliningrad, Russia. (Unknown)
Responsible Party: Principal Investigator, Stepanova Yulia Aleksandrovna, Clinical Professor, National Research Center of Surgery, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: q9ics7t8
Record Dates: First submitted 2019-02-22; First posted 2019-02-28 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2019-02

CONDITIONS: Arrhythmias, Cardiac; Cardiovascular Diseases; Postoperative Atrial Fibrillation; Myocardial Ischemia
Keywords: Bipolar radiofrequency ablation; Atrial Fibrillation New Onset; CABG; Coronary artery disease; Postoperative atrial fibrillation
MeSH Terms: conditions — Arrhythmias, Cardiac; Cardiovascular Diseases; Myocardial Ischemia; Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional CABG (Active Comparator): Coronary artery bypass grafting (CABG) treatment (CABG group,n=70)
  Interventions: Procedure: Conventional CABG
- CABG+ PVI (Active Comparator): CABG + prophylactic epicardial bipolar radiofreaquency pulmonary veins isolation (CABG +PVI group, n=70)
  Interventions: Procedure: CABG+ PVI
- CABG+ PVI+amiodarone (Active Comparator): CABG+ prophylactic epicardial bipolar radiofreaquency pulmonary veins isolation + amiodarone (CABG +PVI+ class III antiarrhythmic drug- amiodarone, group, n=70)
  Interventions: Procedure: CABG+ PVI+amiodarone
- CABG+amiodarone (Active Comparator): CABG+class III antiarrhythmic drug- amiodarone, group, n=70
  Interventions: Procedure: CABG+amiodarone

INTERVENTIONS:
Procedure: Conventional CABG — Coronary artery bypass grafting
  Arms: Conventional CABG
Procedure: CABG+ PVI — CABG+ prophylactic epicardial bipolar radiofrequency isolation of the pulmonary veins
  Arms: CABG+ PVI
Procedure: CABG+ PVI+amiodarone — CABG+PVI+amiodarone (CABG+RFA + class III antiarrhythmic drug- amiodarone)
  Arms: CABG+ PVI+amiodarone
Procedure: CABG+amiodarone
  Arms: CABG+amiodarone

SUMMARY:
To compare prophylactic strategies of atrial fibrillation in patients with CAD and without AF.

DETAILED DESCRIPTION:
Prospective, multicenter, randomized trial, intended to compare three prophylactic strategies of atrial fibrillation in patients with coronary artery disease and without history of atrial fibrillation.

The study includes 4 groups of patients:

Group I (conventional CABG)

Group II (CABG + pulmonary veins isolation). Concomitant CABG and epicardial bipolar radiofrequency pulmonary veins isolation.

Group III (CABG+ pulmonary veins isolation + amiodarone). Concomitant CABG and epicardial bipolar radiofrequency pulmonary veins ablation with administration of amiodarone in postoperative periode.

Group IV (CABG+ amiodarone). Conventional CABG with administration of amiodarone in postoperative periode.

ELIGIBILITY:
Inclusion Criteria:

* patients must have signed an informed consent.
* patients had indications for two or more coronary arteries to be bypassed
* no history of AF

Exclusion Criteria:

* acute coronary syndrome
* previous CABG.
* a significant decrease in the contractile function of the heart (EF <40%)
* significant heart valve disease requiring surgical repair
* long-standing persistent, persistent, or paroxysmal forms of atrial fibrillation
* respiratory failure
* left ventricular aneurysm requiring surgical correction
* chronic renal failure (≤60 mL/min/1⋅73 m2)
* chronic diseases that make a significant contribution to the prognosis of life (e.g. oncology)
* participation in other clinical trials

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2016-09-01; Primary Completion 2016-12-01 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation after CABG | Through study completion, an average of 1 year
Major cardiovascular and cerebral events (MACCE), including death, nonfatal myocardial infarction, repeated revascularization using PCI or CABG, transitory ischemic attack (TIA) or stroke. | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Sinus rhythm at the time of discharge of the patient from the hospital | Through study completion, an average of 1 year
Duration of mechanical ventilation | Through study completion, an average of 1 year
Incidence of implantation of the pacemaker | Through study completion, an average of 1 year
Volume of intraoperative bleeding | Through study completion, an average of 1 year
Time of CBP | Through study completion, an average of 1 year
Time clamping of the aorta | Through study completion, an average of 1 year
Length of stay in the intensive care unit | Through study completion, an average of 1 year
Duration of the hospitalization | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Amiran Sh. Revishvili, Study Chair — A.V. Vishnevsky National Medical Research Center of Surgery. Moscow. Russian Federation.
Locations (2):
- Russia (2):
  - Federal Centre of High Medical Technologies of the RF Ministry of Public Health, Kaliningrad, Russia., Kaliningrad
  - A.V. Vishnevsky National Medical Research Center of Surgery., Moscow